CLINICAL TRIAL: NCT06871904
Title: Exploring the Fibrosis-Modulating Potential of Metformin and Pirfenidone in Oral Submucous Fibrosis: Molecular Mechanisms to Clinical Applications
Brief Title: Fibrosis-Modulating Effects of Metformin and Pirfenidone in Oral Submucous Fibrosis
Acronym: "FIBR-MET-PF"
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ziauddin University (Other)
Collaborators: University of Karachi (Other)
Responsible Party: Principal Investigator, Dr. Afifa Razi, Professor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9840125ARMM; Ethical Review Committee (Other: Ziauddin Univeristy)
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Oral Submucous Fibrosis
Keywords: Oral submucous fibrosis; Fibrosis Modulation; Metformin; Pirfenidone; Exosome secretion; Molecular Pathway; LCMS; Clinical Trial; Exosome Protein Profiling
MeSH Terms: conditions — Oral Submucous Fibrosis | interventions — Metformin; Tablets; pirfenidone; Vitamin E

STUDY DESIGN:
Intervention Model Description: Clinical Trial :All groups will undergo a 24-week intervention phase. The groups will be divided according to the treatment regime.
  Group 1 Control (Supportive Care): Beclomethasone mouthwash three times + Capsule vitamin E 400mg daily.
  Group 2 (Metformin + Supportive Care): Metformin: 500 mg twice daily + Beclomethasone mouthwash three times + Capsule vitamin E 400mg daily.
  Group 3 (Pirfenidone + Supportive Care): Pirfenidone: twice 200 mg daily + Beclomethasone mouthwash three times + Capsule vitamin E 400mg daily.
  Each group will be advised to refrain from spicy ingredients and cease eating pan, chalia or gutkha. All groups will be instructed to perform a mouth-opening stick exercise twice daily, alternating sides, holding the stick for 10 minutes on each side, with a 10-minute rest in between.Clinical evaluations will be conducted every 4 weeks
Who Masked: Participant
Masking Description: double-blind intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Beclomaethasone and Vitamin E (Active Comparator): Group 1 Control (Supportive Care): Beclomethasone mouthwash three times + Capsule vitamin E 400mg daily.
  Interventions: Drug: Beclomaethasone and Vitamin E
- Metformin + Supportive Care (Experimental): Group 2 (Metformin + Supportive Care): Metformin: 500 mg twice daily + Beclomethasone mouthwash three times + Capsule vitamin E 400mg daily.
  Interventions: Drug: Metformin Hydrochloride 500Mg Tablet; Drug: Beclomaethasone and Vitamin E
- Pirfenidone + Supportive Care (Experimental): Group 3 (Pirfenidone + Supportive Care): Pirfenidone: 200 mg twice daily + Beclomethasone mouthwash three times + Capsule vitamin E 400mg daily.
  Interventions: Drug: Pirfenidone (PFD); Drug: Beclomaethasone and Vitamin E

INTERVENTIONS:
Drug: Metformin Hydrochloride 500Mg Tablet — Metformin 500 mg is being tested for its potential role in treating oral submucous fibrosis (OSF) due to its antifibrotic and anti-inflammatory effects. This intervention will be administered orally at a dose of 500 mg twice daily (OD) for a specified 6 months treatment period for Group 2 .
  Metformin activates AMPK (AMP-activated protein kinase), which inhibits TGF-β signaling and collagen deposition, reducing fibrosis and inflammation.
  Distinction from Other Arms: Unlike Pirfenidone, which directly targets profibrotic cytokines, Metformin modulates metabolic pathways to exert antifibrotic effects. The Control Group will receive supportive care for OSF.
  Other Names: Glucophage
  Arms: Metformin + Supportive Care
Drug: Pirfenidone (PFD) — Pirfenidone 200 mg (Pirfibet by Mactor Pharma, Pakistan) is an antifibrotic drug being tested for its potential role in treating oral submucous fibrosis (OSF). This intervention will be administered orally at a dose of 200 mg, twice daily for a specified treatment period which will be 6 months for Group 3 .
  Pirfenidone modulates fibrotic pathways by inhibiting TGF-β and collagen synthesis, reducing fibrosis progression.
  Distinction from Other Arms: Unlike Metformin, which has antifibrotic effects via AMPK activation, Pirfenidone specifically targets profibrotic cytokines. The Control Group will receive either a supportive care for OSF
  Other Names: Pirfibet
  Arms: Pirfenidone + Supportive Care
Drug: Beclomaethasone and Vitamin E — The Supportive Care Group will receive Beclomethasone mouthwash (three times daily) and Vitamin E 400 mg (once daily) as part of supportive care for oral submucous fibrosis . This intervention serves as a comparison group to evaluate the efficacy of Metformin and Pirfenidone.
  Beclomethasone is a topical corticosteroid that reduces inflammation and provides symptomatic relief in OSF.
  Vitamin E is an antioxidant that may help reduce oxidative stress and improve tissue healing.
  Distinction from Other Arms:
  Unlike Pirfenidone and Metformin, which target fibrosis at the molecular level, Beclomethasone + Vitamin E primarily focus on symptom relief.
  This arm will serve as an active comparator to determine whether the antifibrotic effects of Metformin and Pirfenidone provide superior therapeutic benefits.
  Other Names: Beclamethasone; Vitamin E

SUMMARY:
The goal of this clinical trial is to learn if metformin and antifibrotic drugs (pirfenidone) can modulate fibrosis and improve treatment outcomes in patients with oral submucous fibrosis (OSF). The study also aims to investigate the molecular mechanisms underlying their effects on exosome secretion and protein expression.

The main questions it aims to answer are:

Do metformin and antifibrotic drugs alter exosome secretion and biological activity in OSF cell lines? What molecular pathways are influenced by these drugs in modulating fibrosis? Does treatment with metformin and antifibrotic drugs improve clinical outcomes in OSF patients? Researchers will compare metformin and antifibrotic drug treatment groups to a control group to see if these drugs lead to significant changes in fibrosis-related exosomal protein expression and clinical improvement in OSF patients.

Participants will :

Undergo in vitro experiments on OSF cell lines to analyze drug effects using qPCR, Western Blot, and LCMS for protein profiling.

Participate in a randomized, double-blind clinical trial where they receive metformin, antifibrotic drugs, or a placebo.

Undergo clinical evaluations and laboratory tests to assess treatment efficacy. This study aims to develop an affordable and effective fibrosis-targeted therapy for OSF by repurposing metformin, potentially improving patient outcomes and reducing the risk of malignant transformation.

DETAILED DESCRIPTION:
Oral submucous fibrosis stands as a persistent inflammatory and potentially malignant condition affecting the oral cavity, marked by progressive fibrosis of the oral mucosa. Existing therapies, such as corticosteroids, are costly and merely treat the symptoms without addressing the molecular pathways that cause fibrosis, which results in limited efficacy, relapse, and side effects. Given the financial constraints of affected communities, there is a desperate need for affordable and accessible treatments. This research project aims to investigate the effects of metformin and antifibrotic drugs on the secretion and biological activity of exosomes in oral submucous fibrosis (OSF) cell lines. The study will explore how these treatments impact morphological changes, exosomal gene expression, and protein profiles in OSF cell lines compared to control and vehicle-controlled groups. Additionally, the project will identify molecular pathways influenced by metformin and antifibrotic drugs, with a focus on their modulation of exosomal protein content and functional profiles. The clinical relevance of exosomal protein profiles in OSF treatment, particularly through the repurposing of metformin, will also be evaluated. Methodologically, the study involves in vitro experiments on OSF cell lines, employing techniques such as qPCR, Western Blot, and Liquid Chromatography-Mass Spectrometry (LCMS) for protein profiling, alongside a clinical trial to assess therapeutic efficacy.

The project is structured around several key objectives:

1. Impact Assessment: Evaluate how metformin and antifibrotic drugs affect exosome secretion and activity in OSF cell lines.
2. Morphological and Gene Expression Analysis: Analyze morphological changes and exosomal gene expression profiles in OSF cell lines post-treatment compared to control groups.
3. Molecular Pathways: Identify and analyze the molecular pathways modulated by metformin and antifibrotic drugs that influence exosomal protein content and functions.
4. Exosome Characterization: Characterize exosomes isolated from different treatment groups using advanced techniques such as dynamic light scattering (DLS), scanning electron microscopy (SEM), Western Blot (WB) and Liquid Chromatography-Mass Spectrometry (LCMS).
5. Clinical Relevance: Explore the potential clinical applications of the exosomal protein profiles for OSF treatment, focusing on the repurposing of metformin.
6. Methodology: The study includes both in vitro and clinical components, with the in vitro studies involving dose-response experiments, microscopy, gene expression analysis, and exosome isolation and characterization. The clinical trial will assess the efficacy of metformin and antifibrotic drugs in patients with OSF through randomized double-blind controlled trials.

This research has the potential to uncover new therapeutic strategies for OSF, particularly through the repurposing of metformin, which could lead to better clinical outcomes for patients suffering from this precancerous condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with OSF having fibrous bands
2. Patients with limited mouth opening due to OSF in Stage 2 and Stage 3
3. Patients who have not received any treatment for OSF in the previous three months
4. Patients with habits of pan, Chalia, Gutkha
5. The age group between 18 and 45 years

Exclusion Criteria:

1. Patients presenting with OSCC
2. Patients with limited mouth opening due to impaction of the third molar
3. Patients with limited mouth opening due to temporomandibular joint disorder
4. Any history of Metformin intolerance or contraindications to its use.
5. Medical conditions (e.g., cardiovascular disease, renal/hepatic impairment) or drug therapy (>6 months) with immunosuppressants, corticosteroids, or antifibrotics.
6. Pregnancy or lactation.
7. Participation in other clinical trials concurrently.
8. Inability / unwilling to provide informed written consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Exosome Secretion and Characterization in OSF Cell Lines | 24, 48, and 72 hours post-treatment
  This outcome evaluates the effect of Metformin and Pirfenidone on exosome secretion and size distribution in OSF cell lines. Exosomes will be isolated and characterized using Scanning Electron Microscopy (SEM) and Dynamic Light Scattering (DLS) to assess morphological changes, size, and concentration differences across treatment groups.
Changes in Fibrosis-Related Gene Expression in OSF Cell Lines | 24 and 48 hours post-treatment
  This outcome assesses the effect of Metformin and Pirfenidone on fibrosis-related gene expression (TGF-β, Collagen 1A1, α-SMA) in OSF cell lines. Changes will be analyzed using quantitative PCR (qPCR).
Reduction in Fibrosis Severity in OSF Patients | Baseline, 4 weeks, 8 weeks, and 12 weeks, 16 weeks, 20 weeks and 24 weeks
  This outcome measures clinical improvement in Oral Submucous Fibrosis (OSF) patients treated with Metformin, Pirfenidone, or Supportive Care (Beclomethasone + Vitamin E). Severity will be assessed using the Burning Mouth Index by verbal numeric rating scale (0-10) at baseline and every 4 weeks during the trial and Interincisal Mouth Opening (IMO).
Change in TGF-β and Collagen Levels in Exosomes from OSF Cell Lines | 24, 48, and 72 hours post-treatment
  This outcome assesses whether Metformin and Pirfenidone reduce fibrosis-related molecular markers (TGF-β and Collagen) in exosomes isolated from OSF cell lines. Exosomal protein levels will be analyzed using Western Blot and Liquid Chromatography-Mass Spectrometry (LCMS) to determine drug-induced changes in fibrosis-related pathways.

SECONDARY OUTCOMES:
Morphological Changes in OSF Cell Lines Post-Treatment | 24, 48, and 72 hours post-treatment
  This outcome evaluates the morphological alterations in OSF cell lines following treatment with Metformin and Pirfenidone. Changes in cell shape, size, and fibrosis-associated structural modifications will be assessed using Scanning Electron Microscopy (SEM).
Size and Distribution of Exosomes in OSF Cell Lines | 24, 48, and 72 hours post-treatment
  This outcome measures changes in exosome size, distribution, and concentration after treatment with Metformin and Pirfenidone. Characterization will be performed using Dynamic Light Scattering (DLS) and Scanning Electron Microscopy (SEM).
Functional Impact of Treated OSF cells | 24, 48, 72 and 96 hours post- treatment
  This outcome evaluates whether Metformin- and Pirfenidone-treated OSF cell lines, as compared to control untreated OSF cells, influence fibroblast migration and proliferation. Cell behavior will be assessed through Scratch migration and proliferation assays to determine functional effects.
Safety and Viability of OSF Cell Lines Post-Treatment | 24, 48, and 72 hours post-treatment
  This outcome measures the cytotoxicity and cell viability of OSF cell lines following treatment with Metformin and Pirfenidone. MTT assay will be used to assess potential toxic effects of the drugs at different concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because this study involves in vitro experiments on OSF cell lines and does not include individual patient data. Additionally, for the clinical trial component, data privacy regulations and ethical considerations prevent the sharing of participant-specific data

REFERENCES:
- [Background] Wang L, Zhong NN, Wang X, Peng B, Chen Z, Wei L, Li B, Li Y, Cheng Y. Metformin Attenuates TGF-beta1-Induced Fibrosis in Salivary Gland: A Preliminary Study. Int J Mol Sci. 2023 Nov 13;24(22):16260. doi: 10.3390/ijms242216260. PMID 38003450
- [Background] Huh JY, Lee JH, Song JW. Efficacy and safety of combination therapy with pirfenidone and nintedanib in patients with idiopathic pulmonary fibrosis. Front Pharmacol. 2023 Dec 12;14:1301923. doi: 10.3389/fphar.2023.1301923. eCollection 2023. PMID 38192410
- [Background] Chen X, Xie H, Guo J. Drug treatment for oral submucous fibrosis: an update. BMC Oral Health. 2023 Oct 12;23(1):748. doi: 10.1186/s12903-023-03488-9. PMID 37828490
- [Background] Ahmadpour F, Rasouli HR, Talebi S, Golchin D, Esmailinejad MR, Razie A. Effects of exosomes derived from fibroblast cells on skin wound healing in Wistar rats. Burns. 2023 Sep;49(6):1372-1381. doi: 10.1016/j.burns.2023.02.003. Epub 2023 Feb 14. PMID 36828692
- [Background] Abbasi-Malati Z, Azizi SG, Milani SZ, Serej ZA, Mardi N, Amiri Z, Sanaat Z, Rahbarghazi R. Tumorigenic and tumoricidal properties of exosomes in cancers; a forward look. Cell Commun Signal. 2024 Feb 15;22(1):130. doi: 10.1186/s12964-024-01510-3. PMID 38360641
- [Background] Abbasi R, Nejati V, Rezaie J. Exosomes biogenesis was increased in metformin-treated human ovary cancer cells; possibly to mediate resistance. Cancer Cell Int. 2024 Apr 16;24(1):137. doi: 10.1186/s12935-024-03312-6. PMID 38627767